CLINICAL TRIAL: NCT01862822
Title: Position of Children During Urine Collection: Evaluation Study
Acronym: PUCES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: I11 016
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2016-08

CONDITIONS: Urinary Infection
Keywords: Paediatrics; Urinary tract infection; Urine collection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- upright position (Experimental): Upright position during urine bag collection
  Interventions: Other: upright position
- usual position (No Intervention)

INTERVENTIONS:
Other: upright position
  Other Names: the impact of an upright position on the number of contaminated urine cultures during urine bag collection
  Arms: upright position

SUMMARY:
Urinary tract infection (UTI) is a frequently suspected cause of fever in young children, justifying urine cultures. Sampling procedures are decisive for the reliability of UTI diagnosis. Even though official guidelines recommend clean catch method, catheterization or suprapubic aspiration, urine bag collection remains widely used. In our experience, the rate of contaminated bag-obtained cultures reaches 30.2 %. In a recent study, the investigators have noticed that the rate of contaminated urine cultures was lower when children were kept in an upright position at the time of urine collection. The upright position could explain this decrease, perineum being less in contact with urine. These results are borderline significant, the investigators would like to confirm them with a specific study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 - 36 months
* Non-toilet-trained children
* Indication to bag urine collection with the following criteria :
* fever ≥ 38.5 °C
* unexplained fever
* and at least 1 of the following criteria for girls and uncircumcised boys, at least 2 criteria for circumcised boys :
* age ≤ 12 months
* fever ≥ 48 hours
* poorly tolerated fever (chills ± cyanosis ± pronounced weakness…)
* preceding episode of tract urine infection

Exclusion Criteria:

* Parents opposed to the participation of their children in the study
* Diarrhea
* Current antibiotic treatment or during the 8 preceding days of the urine collection
* Genitals / perineal anomaly

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 803 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of polybacterial urine analysis in each group | 1 hour

SECONDARY OUTCOMES:
The failure rate in upright position in private practice | 1 hour.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, Limoges, France

REFERENCES:
- [Result] Bahans C, Dallocchio A, Tran A, Dubos F, Soto B, Schoder G, Blanc P, Messager V, Demonchy D, Labrunie A, Garnier F, Guigonis V. The position during urine sample collection from young precontinent children through a bag does not limit contamination rates: Results from a randomized controlled trial: Does infant position influence quality of urine collection? Arch Pediatr. 2022 Jul;29(5):359-363. doi: 10.1016/j.arcped.2022.03.007. Epub 2022 May 2. PMID 35513967